CLINICAL TRIAL: NCT07123337
Title: Serum 25-Hydroxyvitamin D and Neurological Disability in Multiple Sclerosis: A Cross-Sectional Study From the Mediterranean Epidemiological Frontier
Brief Title: Serum 25-Hydroxyvitamin D and Neurological Disability in Multiple Sclerosis
Acronym: EDSS
Status: Completed | Type: Observational
Sponsor: University of Zintan (Other)
Responsible Party: Sponsor
Other Study IDs: ZFM/2023/MS-01
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-04

CONDITIONS: Multiple Sclerosis
Keywords: EDSS; MS
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Vitamin D is hypothesized to play a role in the immunopathology and progression of multiple sclerosis (MS), yet its association with neurological disability remains uncertain, particularly in North African populations.We conducted a cross-sectional study involving 369 adult MS patients across two tertiary neurology centers in Western Libya. Serum 25-hydroxyvitamin D [25(OH)D] levels and Expanded Disability Status Scale (EDSS) scores were collected. Pearson correlation, ANOVA, and multivariable linear regression were used to assess associations between vitamin D and disability, adjusting for age, BMI, disease duration, and physical activity. Missing data and outliers were handled systematically using validated R and Python workflows.

ELIGIBILITY:
Inclusion Criteria:

* Libyan nationals.
* aged 18 years or older.
* diagnosis of MS based on the 2017 revised McDonald criteria.
* capable of providing informed consent.
* had complete clinical, demographic, and biochemical data.

Exclusion Criteria:

* presence of other neurological disorders that could mimic MS (e.g., neuromyelitis optica spectrum disorder or Lyme disease).
* missing or incomplete medical records.
* pregnancy or lactation.
* extreme psychiatric or cognitive impairment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Libyan male and females between 18 to 70 years diagnosed as MS
Sampling Method: Non-Probability Sample
Enrollment: 369 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
EDSS | 24 months
  interaction between levels of Vit D and EDSS
Serum 25-Hydroxyvitamin D | 24 months
  levels of Vit D

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine zintan university, Tripoli, Tripoli, Libya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vasileiou ES, Hu C, Bernstein CN, Lublin F, Wolinsky JS, Cutter GR, Sotirchos ES, Kowalec K, Salter A, Saidha S, Mowry EM, Calabresi PA, Marrie RA, Fitzgerald KC. Association of Vitamin D Polygenic Risk Scores and Disease Outcome in People With Multiple Sclerosis. Neurol Neuroimmunol Neuroinflamm. 2022 Nov 23;10(1):e200062. doi: 10.1212/NXI.0000000000200062. Print 2023 Jan. PMID 36418179
- [Background] Gill A, Orji C, Reghefaoui M, Peresuodei TS, Thota P, Saavedra Palacios MS, Arcia Franchini AP. The Effectiveness of Vitamin D Intake in Improving Symptoms and Relapses of Multiple Sclerosis: A Systematic Review. Cureus. 2024 Sep 3;16(9):e68565. doi: 10.7759/cureus.68565. eCollection 2024 Sep. PMID 39364460
- [Background] Hanaei S, Sahraian MA, Mohammadifar M, Ramagopalan SV, Ghajarzadeh M. Effect of Vitamin D Supplements on Relapse Rate and Expanded Disability Status Scale (EDSS) in Multiple Sclerosis (MS): A Systematic Review and Meta-Analysis. Int J Prev Med. 2021 May 15;12:42. doi: 10.4103/ijpvm.IJPVM_208_20. eCollection 2021. PMID 34211673